CLINICAL TRIAL: NCT05539859
Title: Efficacy and Safety of NeuroEndoscopic Surgery for IntraCerebral Hemorrhage: a Randomised, Controlled, Open-label, Blinded Endpoint Trial
Brief Title: Efficacy and Safety of NeuroEndoscopic Surgery for IntraCerebral Hemorrhage
Acronym: NESICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Rong Hu, MD, Director of Department of Neurosurgery, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (A)KY2022103
Record Dates: First submitted 2022-09-04; First posted 2022-09-14 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-03

CONDITIONS: Intracerebral Hemorrhage Basal Ganglia
Keywords: Intracerebral hemorrhage; NeuroEndoscopic Surgery
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Endoscopy; Practice Management, Medical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Endoscopic surgery
  Interventions: Procedure: Endoscopic surgery
- Control Arm (Active Comparator): Medical management
  Interventions: Other: Medical management

INTERVENTIONS:
Procedure: Endoscopic surgery — Subjects will receive surgical hematoma evacuation using neuroendoscope, followed by medical management
  Arms: Experimental Arm
Other: Medical management — Subjects will initially receive the standard medical therapies for the treatment of intracerebral hemorrhage, according to the latest available guideline.
  Arms: Control Arm

SUMMARY:
To compare the efficacy and safety of neuroendoscopic hematoma removal and standard conservative treatment for patients with spontaneous supratentorial deep intracerebral hemorrhage.

DETAILED DESCRIPTION:
Neuroendoscopic treatment of spontaneous intracerebral hemorrhage (ICH) is more and more widely used, but multi-center clinical study on the efficacy and safety of neuroendoscopic treatment of ICH is relatively small. Based on the lack of sufficient clinical evidence, the investigators plan to conduct a prospective, multicenter, randomized controlled clinical trial to investigate the safety and efficacy of neuroendoscopy in the treatment of spontaneous cerebral parenchymal hemorrhage, so as to provide evidence-based medical evidence for endoscopic minimally invasive treatment of cerebral hemorrhage and its application.The aim of trial was to determine whether the endoscopic surgery could achieve the benefits of clot evacuation and improve functional outcome at 180 days after ICH without procedure-related safety events or additional brain injury beyond the risks associated with standard care

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, either sex.
2. Time from onset to the first diagnostic CT within 24 hours (for those without bystanders and with unknown onset time, use the last known time the patient was in good condition)
3. Deep (external capsule, putamen, internal capsule, caudate nucleus) supratentorial cerebral hemorrhage with a hematoma volume ≥ 25 ml.
4. Stability of the hematoma determined by two CT scans at different times after onset. If the hematoma enlarges 5ml then the stability of the hematoma can be detected by CT again after 6 hours until the randomization time window is closed.
5. Pre-randomization GCS score of 5-14 and/or NIHSS score of ≥6.
6. Pre-onset Modified Rankin Scale (mRS) score 0 or 1.
7. Blood pressure recorded 6 hours prior to randomization consistently controlled at 180 mmHg or less.
8. Randomization completed within 24 hours after the first diagnostic CT, and surgical intervention should be performed as soon as possible, no later than 6 hours after randomization, that is to say, surgery should be performed no later than 54 hours after onset.
9. Informed and voluntarily signed informed consent by the patient or family.

Exclusion Criteria:

1. Hemorrhage clinically diagnosed as a result of cerebral aneurysm, cerebrovascular malformation, moyamoya disease, traumatic brain injury, brain tumor, hemorrhagic transformation of a large cerebral infarct, coagulation dysfunction.
2. Lobar hemorrhages, thalamic hemorrhages, primary ventricular hemorrhages, cerebellum hemorrhages and brain stem hemorrhages.
3. Hematoma involving the midbrain, with dilated or unresponsive pupils.
4. Hematoma producing life-threatening occupying effects (e.g., CT showing midline deviation of more than 1 cm, loss of cisterna ambiens) or patients who are extremely unstable and unfit for enrollment.
5. Platelet count <100×10^9/L, international normalized ratio (INR) >1.4.
6. Hematoma extension to ventricle and completely blocked the third or fourth ventricle.
7. Recent history of cerebral hemorrhage (less than 1 year).
8. Severe hepatic impairment with ALT 3 times the upper limit of normal, or AST 3 times the upper limit of normal. Severe renal insufficiency with glomerular filtration rate less than 30 ml/min/1.73 m2.
9. Blood pressure not effectively controlled to less than 180 mmHg despite aggressive antihypertensive therapy prior to randomization.
10. Patients with severe advanced cognitive impairment (e.g. AD) or psychiatric disorders who are unable to complete the follow-up program as required.
11. Comorbid other serious diseases such as respiratory, circulatory, digestive, urological, endocrine, immune and hematologic disorders.
12. Pregnant or lactating women, or those who expect to become pregnant within one year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with Modified Rankin Scale (mRS) score 0-3 | 180 days
  Functional outcome (comparing the intervention group to the control), assessed with the modified Rankin Scale (mRS) at 6 months.The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death.
Safety outcome | 180 days
  All cause mortality from onset to 180 days

SECONDARY OUTCOMES:
Glasgow Outcome Scale Extended (GOS-E) | 30 days.
  GOS-E subdivides the categories of severe and moderate disability and good recovery using a scale of 1 to 8 where 1 = death, 2 = vegetative state, 3 = lower severe disability, 4 = upper severe disability, 5 = lower moderate disability, 6 = upper moderate disability, 7 = lower good recovery, and 8 = upper good recovery. Structured telephone interviews have been developed and validated for the GOS-E and these questions were incorporated into the follow-up survey. GOS-E was dichotomized into unfavorable (1 to 4) and favorable (5 to 8) outcomes.
Glasgow Outcome Scale Extended (GOS-E) | 90 days.
  GOS-E subdivides the categories of severe and moderate disability and good recovery using a scale of 1 to 8 where 1 = death, 2 = vegetative state, 3 = lower severe disability, 4 = upper severe disability, 5 = lower moderate disability, 6 = upper moderate disability, 7 = lower good recovery, and 8 = upper good recovery. Structured telephone interviews have been developed and validated for the GOS-E and these questions were incorporated into the follow-up survey. GOS-E was dichotomized into unfavorable (1 to 4) and favorable (5 to 8) outcomes.
Glasgow Outcome Scale Extended (GOS-E) | 180 days.
  GOS-E subdivides the categories of severe and moderate disability and good recovery using a scale of 1 to 8 where 1 = death, 2 = vegetative state, 3 = lower severe disability, 4 = upper severe disability, 5 = lower moderate disability, 6 = upper moderate disability, 7 = lower good recovery, and 8 = upper good recovery. Structured telephone interviews have been developed and validated for the GOS-E and these questions were incorporated into the follow-up survey. GOS-E was dichotomized into unfavorable (1 to 4) and favorable (5 to 8) outcomes.
Modified Rankin Scale (mRS) Score | 30 days.
  The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death.
Modified Rankin Scale (mRS) Score | 90 days .
  The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death.
Survival rate | 30 days.
  comparing the intervention group to the control
Survival rate | 90 days.
  comparing the intervention group to the control
Assessment of cognitive function with Mini-Mental State Examination (MMSE) | 30 days.
  The MMSE is a screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function.
Assessment of cognitive function with Mini-Mental State Examination (MMSE) | 90 days.
  The MMSE is a screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function.
Assessment of cognitive function with Mini-Mental State Examination (MMSE) | 180 days.
  The MMSE is a screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function.
Quality of life measured with the 5-level EQ-5D (EQ-5D-5L) | 30 days.
  The EQ-5D-5L is a standard measure of health-related quality of life.EQ-5D-5L consists of two components: a health state profile and a visual analog scale (VAS). EQ-5D health state profile comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The 5D-5L systems are converted into a single index utility score between 0 to 1, where a higher score indicates a better health state. The VAS records the participant's health on a 0-100 mm VAS scale, with 0 indicating "the worst health you can imagine" and 100 indicating "the best health you can imagine". Higher scores of EQ VAS indicate better health.
Quality of life measured with the 5-level EQ-5D (EQ-5D-5L) | 90 days.
  The EQ-5D-5L is a standard measure of health-related quality of life.EQ-5D-5L consists of two components: a health state profile and a visual analog scale (VAS). EQ-5D health state profile comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The 5D-5L systems are converted into a single index utility score between 0 to 1, where a higher score indicates a better health state. The VAS records the participant's health on a 0-100 mm VAS scale, with 0 indicating "the worst health you can imagine" and 100 indicating "the best health you can imagine". Higher scores of EQ VAS indicate better health.
Quality of life measured with the 5-level EQ-5D (EQ-5D-5L) | 180 days.
  The EQ-5D-5L is a standard measure of health-related quality of life.EQ-5D-5L consists of two components: a health state profile and a visual analog scale (VAS). EQ-5D health state profile comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The 5D-5L systems are converted into a single index utility score between 0 to 1, where a higher score indicates a better health state. The VAS records the participant's health on a 0-100 mm VAS scale, with 0 indicating "the worst health you can imagine" and 100 indicating "the best health you can imagine". Higher scores of EQ VAS indicate better health.
Length of ICU | Number of days from admission, up to 180 days
  Duration of stay in the ICU
Length of hospitalization | Number of days from admission to discharge, up to 180 days
  Duration of stay in the hospital
In-hospital cost | Number of days from admission to discharge, up to 180 days
  all medical cost during the in-hospital period

CONTACTS AND LOCATIONS:
Overall Officials: Rong Hu, MD, Study Chair — PLA Army Medical University
Locations (4):
- China (4):
  - chongqing Emergency Medical Center, Chongqing, Chongqing Municipality
  - Xiang Yang NO.1 Peoples Hospital, Hubei, Hubei
  - Dazhu County People's Hospital, Sichuan, Sichuan
  - Ganzhou city people's Hospita, Ganzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen BM, Ullman N, Muschelli J, Norrving B, Dlugash R, Avadhani R, Awad I, Zuccarello M, Ziai WC, Hanley DF, Thompson RE, Lindgren A; MISTIE and CLEAR Investigators. Relationship of White Matter Lesions with Intracerebral Hemorrhage Expansion and Functional Outcome: MISTIE II and CLEAR III. Neurocrit Care. 2020 Oct;33(2):516-524. doi: 10.1007/s12028-020-00916-4. PMID 32026447
- [Background] de Oliveira Manoel AL. Surgery for spontaneous intracerebral hemorrhage. Crit Care. 2020 Feb 7;24(1):45. doi: 10.1186/s13054-020-2749-2. PMID 32033578
- [Background] Anderson CD, James ML. Survival and independence after intracerebral hemorrhage: Trends and opportunities. Neurology. 2018 Jun 5;90(23):1043-1044. doi: 10.1212/WNL.0000000000005625. Epub 2018 May 4. No abstract available. PMID 29728523
- [Background] Kuo LT, Chen CM, Li CH, Tsai JC, Chiu HC, Liu LC, Tu YK, Huang AP. Early endoscope-assisted hematoma evacuation in patients with supratentorial intracerebral hemorrhage: case selection, surgical technique, and long-term results. Neurosurg Focus. 2011 Apr;30(4):E9. doi: 10.3171/2011.2.FOCUS10313. PMID 21456936
- [Background] Kellner CP, Song R, Pan J, Nistal DA, Scaggiante J, Chartrain AG, Rumsey J, Hom D, Dangayach N, Swarup R, Tuhrim S, Ghatan S, Bederson JB, Mocco J. Long-term functional outcome following minimally invasive endoscopic intracerebral hemorrhage evacuation. J Neurointerv Surg. 2020 May;12(5):489-494. doi: 10.1136/neurintsurg-2019-015528. Epub 2020 Jan 8. PMID 31915207
- [Background] Xu X, Chen X, Li F, Zheng X, Wang Q, Sun G, Zhang J, Xu B. Erratum. Effectiveness of endoscopic surgery for supratentorial hypertensive intracerebral hemorrhage: a comparison with craniotomy. J Neurosurg. 2018 Feb;128(2):649. doi: 10.3171/2017.5.JNS161589a. Epub 2017 Jul 28. No abstract available. PMID 28753114
- [Derived] Wang L, Zhou T, Wang P, Zhang S, Yin Y, Chen L, Duan H, Wu N, Feng H, Hu R. Efficacy and safety of NeuroEndoscopic Surgery for IntraCerebral Hemorrhage: A randomized, controlled, open-label, blinded endpoint trial (NESICH). Int J Stroke. 2024 Jun;19(5):587-592. doi: 10.1177/17474930241232292. Epub 2024 Feb 19. PMID 38291017